CLINICAL TRIAL: NCT06392815
Title: 64Cu-DOTATATE-PET Imaging for Lyme Neuroborreliosis
Brief Title: 64Cu-DOTATATE-PET for Lyme Neuroborreliosis
Acronym: DOTA-LYME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne-Mette Lebech, Consultant, associate professor, MD Dsc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RH8622
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Borrelia Burgdorferi Neuroborreliosis
Keywords: borrelia burgdorferi; Neuroborreliosis; Dotatate PET
MeSH Terms: conditions — Lyme Neuroborreliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroborreliosis (Other): 25 patients with possible or confirmed neuroborreliosis
  Interventions: Diagnostic Test: Cu DOTATATE PET
- controls (Other): 25 patients investigated for neuroborreliosis but with normal CSF examination
  Interventions: Diagnostic Test: Cu DOTATATE PET

INTERVENTIONS:
Diagnostic Test: Cu DOTATATE PET — The primary endpoint of the study is diagnostic performance for detecting LNB by 64Cu-DOTATATE-PET/CT/MRI measured as the difference in uptake between patients with definite LNB and patients without LNB. The primary read-out from 64Cu-DOTATATE-PET/CT/MRI is SUV in CNS and reference organs

SUMMARY:
The aim of the study is to investigate the applicability and performance of 64Cu-DOTATATE PET/CT/MR for diagnosis in patients with Lyme neuroborreliosis (LNB).

In this prospective, observational cohort study with 64Cu-DOTATATE, the investigators wish to include a total of 50 patients clinically suspected of LNB. The investigators will investigate the diagnostic value of 64Cu-DOTATATE-PET comparing clinically suspected and CSF verified LNB patients with clinically suspected patients without CSF verification.

The investigators hypothesize that the information obtained from 64Cu-DOTATATE PET/CT/MRI can improve the diagnostics of LNB as well as that 64Cu-DOTATATE PET/CT/MRI will be able to contribute to the follow-up of patients by adding prognostic information and the risk of persistent symptoms. The application of 64Cu-DOTATATE PET/CT/MRI in the diagnostic work-up of LNB would thus expectedly lead to a more precise diagnosis and risk assessment.

DETAILED DESCRIPTION:
Background

Imaging of neuroinfections is well documented, however with several restrictions due to the heterogeneity of pathogens. Lyme neuroborreliosis (LNB) is a tick-borne infection, caused by Borrelia burgdorferi sensu lato complex (Bb) and among the most prevalent bacterial infections of the nervous system. Due to climatic and environmental changes, the incidence of tickborne diseases is increasing throughout Europe, in Denmark the annual incidence is estimated to 3-4/100,000. Adults mainly manifests as a self-limiting subacute painful meningoradiculitis, lymphocytic meningitis and/or cranial nerve palsy, symptoms of CNS involvement such as acute encephalitis and myelitis are rare. Over time, most cases of Bb infection is thought to be self-resolving, however antibiotics accelerate the process by eradicating the pathogen and reduces the risk of disseminated late infection and persistent symptoms. The response to antibiotics can be slow, but the majority of patients report marked improvement in symptoms after treatment, a proportion of patients, do however report to experience persistent residual symptoms including fatigue, pain or cognitive disturbances and studies have suggested that late diagnosis and the burden of symptoms at time of treatment initiation increases the risk of these symptoms.

If antibiotic treatment is initiated as early as possible, LNB has a very good prognosis, early diagnosis and treatment initiation are therefore of paramount interest.

As no markers in plasma can be used to diagnose or follow LNB, the diagnosis of LNB is based on clinical symptoms in combination with elevated white blood cell count in cerebrospinal fluid (CSF) and the detection of specific Bb intrathecal antibody production. However, Bb serology has several disadvantages in the ability to confirm active disease and monitor disease activity and response to antibiotic treatment. Bb antibodies in CSF are first detectable weeks after onset of the neuroinfection and they may persist for years even after the disease has been well-treated. In addition, symptoms can be unspecific, evolving over time and even mimic other neurological diseases potentially resulting in misdiagnosis, diagnostic delay and reduced patient outcome. The investigators recently reported a median duration of neurological symptoms before first hospital contact of 21 days in a Danish nationwide prospective cohort study of 194 LNB patients included between 2015-2018. Currently, the only way to monitor disease activity - although not ideal - is to to perform a re-lumbar puncture, which is an invasive procedure, not always possible or successful and with risk of post lumbar puncture headache which develops in 10-20% of the patients.

Improving diagnosis, ideally non-invasively, is therefore of great interest and new methods to confirm active disease and monitor the effect of treatment an important field of research which might promote a shift from empirical treatment to personalized medicine with expected improvement in patient outcome.

Non-invasive imaging seems an obvious solution. The investigators have retrospectively studied the value of CT and MRI in diagnosis of LNB and found no value of computerized tomography (CT)-head and limited value of magnetic resonance imaging (MRI)-Brain/Spine. Regarding use of positron emission tomography (PET) the most commonly used ligand for infection and inflammation imaging is the radiolabeled glucose analogue, fluorine-18-fluorodeoxyglucose (18F-FDG). However, 18F-FDG has major limitations including low specificity, as it is taken up by any cell with increased glucose metabolism including but not restricted to leukocytes, macrophages, monocytes, lymphocytes and giant cells. In addition, as the normal brain has high glucose consumption, it is difficult (impossible) to obtain sufficient contrast in LNB as inflammation is primarily in the meninges. Indeed, the investigators have confirmed from cases of LNB that had 18F-FDG-PET could not be used. Due to these limitations, there is an unmet need for other, more specific, targeted radioligands to improve imaging of infectious diseases e.g. LNB and the adjacent inflammatory response.

Macrophages is a potential and promising target for the diagnosing of more specific infections and in particular LNB. Macrophages have anti-inflammatory properties with high phagocytic activity, and they are not only involved in the early immune response but present as long as the infection is active. Macrophage activation can be monitored by the circulating biomarker soluble CD163, the intrathecal inflammation in LNB does not lead to any or only very subtle peripheral measurable changes of normal infectious parameters even with highly active but localized infection as in LNB. As activated macrophages overexpresses somatostatin receptor subtype 2 (sstr2), the activity of macrophages can be visualized by PET imaging targeting sstr2 using the ligand 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetic acid]-d-Phe1,Tyr3-octreotate (DOTATATE). At Rigshospitalet the investigators recently developed 64Cu-DOTATATE with a physical half-life of 12.7 hours (vs. 1 hour) and a 4-fold better theoretical (positron range) spatial resolution compared to existing 68Ga-labeled tracers. These characteristics are a prerequisite. Accordingly, the investigators found in a pre-clinical trial that 64Cu-DOTATATE was able to non-invasively detect and monitor Lyme borreliosis in a murine model of Lyme arthritis and that delayed imaging, later than 3 h and ideally 24 h post injection, was necessary to obtain good target-to-background ratios in images of Bb infection.

In humans, the investigators previously demonstrated that 64Cu-DOTATATE-PET could visualize macrophages in vivo in atherosclerotic, carotid plaques prior to endarterectomy. Gene expression analysis on the excised plagues demonstrated at close correlation between CD163 gene expression and PET tracer uptake confirming that it was indeed macrophages that were visualized.

In this prospective, observational cohort study with 64Cu-DOTATATE, the investigators wish to include a total of 50 patients clinically suspected of LNB. The investigators will investigate the diagnostic value of 64Cu-DOTATATE-PET comparing clinically suspected and CSF verified LNB patients with clinically suspected patients without CSF verification. The investigators further wish to explore if the biomarkers sCD163, NfL, and Tau may contribute to the diagnostics of LNB, and if 64Cu-DOTATATE PE/CT/MRI have a prognostic value by including a follow-up visit 6 months after treatment, comparing patients with persistent symptoms to patients without persistent symptoms. The investigators hypothesize that the information obtained from 64Cu-DOTATATE PET/CT/MRI and the biomarkers sCD163 and NfL can improve the diagnostics of LNB. The investigators also hypothesize that 64Cu-DOTATATE PET/CT/MRI will be able to contribute to the follow-up of patients by adding prognostic information and the risk of persistent symptoms. The application of 64Cu-DOTATATE PET/CT/MRI in the diagnostic work-up of LNB would thus expectedly lead to a more precise diagnosis and risk assessment.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years AND

* Clinical suspicion of LNB AND
* Must be able to read and understand the patient information and to give informed consent -

Exclusion Criteria:

* Pregnancy OR
* Breast-feeding OR
* Concluded antibiotic treatment OR
* Weight more than the maximum weight limit for the PET/CT/MRI bed of the scanner (140 kg) OR
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 64Cu-DOTATATE OR
* Contraindications to MR (check list) -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary | 2,5 years
  Sensitivity and specificity of 64Cu-DOTATATE PET/CT/MR for detection of LNB in patients clinically suspected of LNB using CSF as reference

SECONDARY OUTCOMES:
Secondary | 2,5 years
  Correlation between responders vs. non-responders on 64Cu-DOTATATE PET/CT/MR and outcome at 6 months measured according to 36-item short form survey (SF-36) score and multidimensional fatigue inventoryscore (MFI-20 score). The SF-36 is a set of self reported quality of life measures.Possible scores range from 0 to 100, with higher scores representing better health status. MFI-20 The MFI is a 20-item self-report instrument designed to measure fatigue.Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Lebech, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Anne-Mette Lebech, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided